CLINICAL TRIAL: NCT01187784
Title: Effectiveness of Cognitive-Behavioral Therapy for Children With High-Functioning Autism Spectrum Disorder and Anxiety
Brief Title: Cognitive-Behavioral Therapy for Children With High-Functioning Autism Spectrum Disorder and Anxiety
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Alliant International University (Other)
Collaborators: National Foundation for Autism Research (Unknown); Autism Society of America - San Diego Chapter (Unknown)
Responsible Party: Rebecca McNally Keehn, M.A., Alliant International University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: McNallyKeehn
Record Dates: First submitted 2010-08-23; First posted 2010-08-24 (Estimated); Last update posted 2010-08-24 (Estimated); Status verified 2010-08

CONDITIONS: Autism Spectrum Disorder; Autism; Asperger Syndrome; PDD-NOS
MeSH Terms: conditions — Autism Spectrum Disorder; Autistic Disorder; Asperger Syndrome

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- CBT (Active Comparator): Coping Cat cognitive-behavioral therapy protocol
  Interventions: Behavioral: Coping Cat cognitive-behavioral therapy for anxious youth
- Waitlist Control (No Intervention): Treatment as usual

INTERVENTIONS:
Behavioral: Coping Cat cognitive-behavioral therapy for anxious youth — Manualized, empirically supported CBT treatment for anxious youth
  Arms: CBT

SUMMARY:
Many children and adolescents with autism spectrum disorder (ASD) experience high levels of anxiety which can further inhibit their ability to master developmental tasks such as succeeding in school and developing and maintaining friendships. Despite the need for effective treatments for children with ASD and anxiety, there have been few studies that have addressed this issue. Recently, preliminary evidence has supported the use of cognitive-behavioral therapy (CBT) to treat anxiety disorders in children with ASD.

This study will utilize a CBT treatment program called Coping Cat. Coping Cat has been found to be one of the most effective treatments for typically developing children with anxiety and has also been shown to be effective for treating anxiety in children with other disorders such as physical impairments, selective mutism, and Attention Deficit Hyperactivity Disorder. The investigators goal is to demonstrate that Coping Cat is an effective treatment for children with ASD and anxiety. Finding effective treatments for children with ASD and anxiety could increase adaptive social relationships, decrease stress among families, and prevent the maintenance of anxiety into adulthood.

DETAILED DESCRIPTION:
The purpose of the current study is to evaluate the effectiveness of an empirically-supported, individually-based cognitive-behavioral treatment for anxiety disorders in children with autism spectrum disorder (ASD). Recent research suggests that 47 - 84% of children with ASD experience clinically significant levels of anxiety due to inhibited temperament, physiological hyperarousal, and distinct information processing biases. Despite the clear need for effective treatments for children with ASD and anxiety, there have been few empirical studies. However, a small body of literature has demonstrated growing support for the use of cognitive-behavioral therapy (CBT) to treat anxiety in children with high-functioning ASD. Kendall and Hedtke's Coping Cat cognitive-behavioral therapy program for anxious children will be utilized as the primary intervention. To date, there are no studies that have used this treatment program for anxiety in children with developmental disorders, including ASD. However, Coping Cat has been successfully adapted for children with a variety of co-occurring diagnoses (e.g., physical impairments, selective mutism). Participants in this study will be 20 children aged 7;0 to 14;11 years diagnosed with high-functioning ASD and at least one anxiety disorder (separation anxiety disorder, generalized anxiety disorder, or social phobia). A randomized controlled trial design will be employed. It is hypothesized that participants in the CBT condition will demonstrate a significantly larger reduction in overall levels of anxiety from pre-treatment to post-treatment compared to those in the waitlist (WL) condition and that children who complete the CBT treatment will maintain gains at two-month follow-up.

ELIGIBILITY:
Inclusion Criteria:

* 7 - 14 years
* Diagnosis of an autism spectrum disorder (meets DSM-IV criteria for autism, Asperger syndrome, or Pervasive Developmental Disorder - Not Otherwise Specified (PDD-NOS))
* Clinically significant anxiety (meets DSM-IV criteria for separation anxiety disorder, social phobia, or generalized anxiety disorder)
* IQ > 70
* Primary spoken language: English

Exclusion Criteria:

* IQ < 70
* Comorbid psychotic disorder

Ages: 7 Years to 14 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 22 (Actual)
Dates: Start 2009-05; Primary Completion 2010-08 (Actual); Study Completion 2010-08 (Actual)

PRIMARY OUTCOMES:
Anxiety Disorders Interview Schedule - Child/Parent Version | Post Treatment (16 weeks)
  Scores on parent-administered anxiety diagnostic interview after treatment or waitlist.

SECONDARY OUTCOMES:
Multidimensional Anxiety Scale for Children | Post Treatment (16 weeks)
  Scores on self-report anxiety rating scale after treatment or waitlist.
Spence Children's Anxiety Scale (Child and Parent Versions) | Post Treatment (16 weeks)
  Scores on self-and parent-report anxiety rating scale after treatment or waitlist.

CONTACTS AND LOCATIONS:
Overall Officials: Rebecca McNally Keehn, M.A., Principal Investigator — Alliant International University
Locations (1):
- Alliant International University, San Diego, California, United States

REFERENCES:
- [Derived] McNally Keehn RH, Lincoln AJ, Brown MZ, Chavira DA. The Coping Cat program for children with anxiety and autism spectrum disorder: a pilot randomized controlled trial. J Autism Dev Disord. 2013 Jan;43(1):57-67. doi: 10.1007/s10803-012-1541-9. PMID 22588377